CLINICAL TRIAL: NCT01120444
Title: A Single Center, Open-label, Randomized Study Examining the Glycemic Effects of ID vs SC Bolus Dosing of Insulin Lispro in Patients With Type 1 Diabetes
Brief Title: Study on the Effects on Blood Glucose Following Intradermal and Subcutaneous Dosing of Insulin in Diabetic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Kevin Judge, MD, Becton, Dickinson and Company
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BDT-09-ADC004
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes
Keywords: Diabetes; Insulin; Blood Glucose
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Needles; Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous delivery of insulin (Active Comparator): A bolus dose of insulin will be given subcutaneously just prior to a standardized meal.
  Interventions: Device: Subcutaneous delivery of insulin using Disetronic Accu-Chek Rapid D infusion set
- Intradermal delivery of insulin (Experimental): A bolus dose of insulin will be given intradermally just prior to a standardized meal
  Interventions: Device: BD Research Catheter with 34G x 1.5 mm needle

INTERVENTIONS:
Device: BD Research Catheter with 34G x 1.5 mm needle — bolus injection of insulin given intradermal prior to standardized meal
  Arms: Intradermal delivery of insulin
Device: Subcutaneous delivery of insulin using Disetronic Accu-Chek Rapid D infusion set — bolus delivery of insulin given subcutaneously prior to standardized meal
  Other Names: Disetronic Accu-Chek Rapid D infusion set - 6mm cannula
  Arms: Subcutaneous delivery of insulin

SUMMARY:
The purpose of this study is to compare the effects of bolus delivery of insulin when delivered either intradermally (in the skin) or subcutaneously (under the skin) in diabetics.

DETAILED DESCRIPTION:
Each patient will participate in 10 visits of which the first, Visit 1, is a Screening Visit.

Visit 2 will consist of a brief isoglycemic clamp with a single IV insulin challenge to determine insulin sensitivity. A subsequent test meal and single SC insulin dose (off clamp) will be done to determine the nominal coverage dose of insulin for a mixed meal containing 60g of carbohydrate. This nominal dose will form the basis of insulin bolus dosing for the remainder of the study visits.

For Visits 3-9, patients will come to the institute in the early morning 24 hours prior to the meal test for the application of a Continuous Glucose Monitor (Dexcom Seven Plus™, Dexcom, INC). Subjects will receive standardized meals during the day and their blood glucose will be stabilized overnight to a concentration of 115±15 mg/dL via IV insulin and/or glucose infusions. The next morning the subjects will start the experimental intervention. Immediately prior to standardized meals (2 minutes before eating) the patients will receive insulin by either the ID or SC route, followed by the breakfast (rapidly absorbed carb) meal at time point T0. Meal consumption will occur over a 10 to 15 min time interval. Blood glucose excursions will be observed in the 6 hours thereafter (until T= 360 min). Between hours 6 to 7, BG may be re-stabilized to starting values (115±15 mg/dL) by administration of IV insulin or glucose if necessary. At that time a second insulin injection (same dose as at time point T= -2 minutes) will be given and a second standardized lunch (mixed) meal will be administered. Blood glucose excursions will be followed for an additional 6 hours thereafter (T = 780 minutes)

Conditions for Visits 3-8 will be:

* Condition 1. Individualized Lispro ID dose (nominal dose based on prior insulin sensitivity testing and patient-specific insulin-to-carb ratio) given immediately (2min) prior to a breakfast meal containing predominantly rapidly absorbed carbohydrates (std 60 g CHO; approximately 70:15:15 CHO:protein:fat); a second lunch mixed meal given 7 hours later contains the same total number of carbohydrates (std 60 g mixed) but with a mixed composition between carbohydrate, protein, and fat (ratio approximately 35:25:40).
* Condition 2. Equivalent insulin dose and meal regimen as Condition 1 but given by the SC route.
* Conditions 3 and 4. The meal regimen from Condition 1, with ID and SC doses increased 30% above the nominal dose to simulate inappropriate carb counting.
* Conditions 5 and 6. The meal regimen from Condition 1, with ID and SC doses decreased 30% below the nominal dose to simulate inappropriate carb counting.

In addition during each meal challenge the subject will be maintained on an Animas pump intradermally delivering a combined bolus and basal profile of a placebo (5% dextrose for injection solution) during the study period to evaluate flow biomechanics.

Visit 9 will examine a single earlier dose timing (determined by analysis of the glycemic profile dataset from the prior 8 visits) relative to the two meals for the ID route only, using the optimal target dose from conditions 1 and 2.

Patients will have a final examination, Visit 10, immediately following Visit 9.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients will be included in the trial only if they fulfill all of the inclusion criteria mentioned below:

* Understood and signed informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the patient)
* Type 1 Diabetes mellitus, according to clinical judgment / ADA / WHO-definition (Diabetes Care 2003; 26: 5-20) for at least 1 year.
* Usage of insulin pump therapy or multiple daily injections ("basal-bolus") with carb counting for at least six months
* Age in the range of ≥18 and ≤55 years
* Body mass index (BMI) ≤32 kg/m²
* HbA1c ≤ 8.0% at screening
* Able and willing to adhere to the study procedures for the entire trial period
* Negative test results for hepatitis C antibodies, hepatitis B surface antigen and HIV at screening.

Exclusion Criteria:

Patients will not be permitted to enter the trial, if they fulfill any of the exclusion criteria mentioned below:

* Previous participation in this trial or participation in a clinical trial within 3 months prior to screening examination
* Any symptoms suggestive of, or a diagnosis or treatment for gastroparesis
* Abnormalities in renal function (e.g. serum creatinine >1.2 mg/dl) or judged by the investigator that would pose a problem of clearance of injected insulin
* Proliferative retinopathy or maculopathy that has required acute treatment within the last six months
* Acute and severe illness apart from diabetes mellitus as judged by the investigator
* Abnormalities in the laboratory parameters if judged as clinically significant by the investigator. In particular, patients with GOT/GPT >3x, thrombocyte count <100/nL, INR >1.3, PTT >50 sec.
* Clinically significant abnormalities in the ECG
* Recurrent major hypoglycemia or hypoglycemic unawareness as judged by the investigator
* Lipodystrophy which in the judgment of the investigator would pose a problem in terms of variability of absorption of injected insulin
* Use of systemic corticoids for the last three month prior screening examination or treatment with medication known to interfere with glucose metabolism such as non-selective ß-blockers, or mono amine oxidase (MAO) inhibitors, ACE-inhibitors or thiazides, unless such medical treatment has existed for at least three months and is not changing, prior to screening examination
* Any disease requiring use of anti-coagulants
* Impaired hepatic or renal functions as judged by the investigator Cardiac problems as judged by the investigator
* Uncontrolled hypertension (treated or untreated) as judged by the investigator (RRsyst. >140 mmHg, RRdiast. > 90 mmHg)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation Current addiction to alcohol or substances of abuse as determined by the investigator
* Allergy to plaster/adhesive
* Any other condition that the investigator feels would interfere with trial participation or evaluation of results.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 12-14 hours
  To compare between the ID and SC routes the relative PD times "in-range" (70-180 mg/dL) for glycemic excursions following two types of standardized meals and three dose ranges (optimum dose and +/- 30%).

SECONDARY OUTCOMES:
Insulin levels | 12-14 hours
  To compare the pharmacokinetics of insulin absorption as well as the intra-subject variability for each delivery routes.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil Institute of Research
Locations (1):
- Profil Institute of Clinical Research, Neuss, Germany